CLINICAL TRIAL: NCT00669994
Title: Prospective, Open Label Non-comparative, Multi-center Trial to Evaluate the Efficacy and Safety of Cipro® XR 500 mg Once Daily for 3 Days in Treating Female Patients With Acute, Uncomplicated, Symptomatic Lower Urinary Tract Infections
Brief Title: Trial to Evaluate the Efficacy and Safety of Cipro® XR in Treating Female Patients With Lower Urinary Tract Infections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100546
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Urinary Tract Infection
Keywords: UTI; Urinary Tract Infection
MeSH Terms: conditions — Urinary Tract Infections | interventions — Ciprofloxacin

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Ciprofloxacin

INTERVENTIONS:
Drug: Ciprofloxacin — Cipro XR 500 mg tablets taken once daily

SUMMARY:
This trial evaluated how effective and safe Cipro XR was in treating female patients with signs and symptoms of a lower urinary tract infections. After 3 days of treatment, patients were evaluated to determine if signs/symptoms disappeared and the infecting bacteria was eliminated.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant, non-lactating female outpatients between the ages of 18 - 44 years (inclusive)
* Patients with at least two of the following clinical signs and symptoms of an uUTI:

  * Dysuria
  * Frequency
  * Urgency
  * Suprapubic pain
* Patients with onset of symptoms < 72 hours prior to study entry
* Patients with one positive pre-treatment clean-catch midstream urine culture at enrollment in the study, defined as > 10000 CFU/mL (study drug treatment is permitted prior to the availability of urine culture results)
* Positive leukocyte esterase (LE) (1+ or greater) utilizing a urine dipstick method of analysis
* Patients willing to give written informed consent
* Cultures must be performed on pre-treatment clean-catch midstream urine (MSU) specimens

Exclusion Criteria:

* Males
* Women who are pregnant, nursing, or not using two medically accepted, effective methods of birth control
* Patients with known or suspected hypersensitivity to quinolones
* Patients unable to take oral medication for any reason
* Patients with an asymptomatic bacteriuria
* Patients with complicated UTI, defined as: a clinical syndrome characterized by the development of systemic and local signs and symptoms of fever (> 38.3°C/101°F orally), chills, malaise, flank pain, back pain, or costovertebral angle (CVA) pain or tenderness
* Symptoms as outlined in the inclusion criteria occurring in the presence of a functional or anatomical abnormality of the urinary tract or in the presence of urinary catheterization
* Patients with symptoms of a UTI within the 4 weeks prior to the present episode
* Patients with the onset of symptoms >72 hours prior to study entry
* Patients with three or more episodes of any UTI in the past 12 months
* Patients with evidence of factors predisposing to the development of UTIs, including calculi, stricture, primary renal disease (e.g. polycystic renal disease), or neurogenic bladder
* Patients who received systemic antimicrobial therapy within 48 hours prior to entry
* Patients with a neutrophil count < 1000/mm3, CD4 < 200/mm3 or other conditions associated with significant depression in host defense; HIV testing is not mandatory
* Patients requiring concomitant systemic antibacterial therapy with agents not specified in this protocol
* Patients with a previous history of tendinopathy associated with fluoroquinolones
* Patients diagnosed with a rapidly fatal underlying disease (death expected within six months)
* Patients requiring concomitant use of theophylline
* Patients previously enrolled in this clinical study
* Patients taking an investigational drug in the last 30 days

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2003-07; Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Bacteriologic outcome in patients with UTI caused by S. saprophyticus | 4-11 days post-treatment

SECONDARY OUTCOMES:
Adverse Events Collection | Up to 4-11 days post-treatment
Clinical Response | 4-11 days post-treatment
Incidence of premature terminations | Premature discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (28):
- United States (28):
  - Birmingham, Alabama
  - Pelham, Alabama
  - Phoenix, Arizona
  - Laguna Hills, California
  - Long Beach, California
  - San Diego, California
  - San Luis Obispo, California
  - San Mateo, California
  - Sylmar, California
  - Yorba Linda, California
  - Avon, Connecticut
  - Clearwater, Florida
  - Pembroke Pines, Florida
  - Evansville, Indiana
  - Milford, Massachusetts
  - Royal Oak, Michigan
  - Elizabeth, New Jersey
  - Holmdel, New Jersey
  - Camillus, New York
  - Beaver, Pennsylvania
  - Feasterville, Pennsylvania
  - Hatboro, Pennsylvania
  - Summerville, South Carolina
  - San Antonio, Texas
  - Murray, Utah
  - Salt Lake City, Utah
  - West Jordan, Utah
  - Madison, Wisconsin